CLINICAL TRIAL: NCT05919342
Title: Screening for earlY Heart Failure Diagnosis and Management in Primary Care or at HOme Using Natriuretic Peptides and echocardiographY
Brief Title: Screening for earlY Heart Failure Diagnosis and Management in Primary Care or at HOme Using Natriuretic Peptides and echocardiographY "SYMPHONY-HF"
Acronym: SYMPHONY-HF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other); National Heart Centre Singapore (Other); Karolinska University Hospital (Other); Uppsala University (Other); Montreal Heart Institute (Other); Rigshospitalet, Denmark (Other); University of British Columbia (Other); The Cleveland Clinic (Other); Université de Montréal (Other); AstraZeneca (Industry); Roche Pharma AG (Industry); Us2.ai (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1
Record Dates: First submitted 2023-05-21; First posted 2023-06-26 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Heart Failure; Cardiovascular Diseases
Keywords: Screening; Biomarker; NT-proBNP; Echocardiography; Community; Registry
MeSH Terms: conditions — Heart Failure; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: After agreeing to consent, patients will be randomised 1:1 to one of two arms; a "Routine care arm" in which patients will undergo routine care or a 2. "Investigational arm" - patients in this arm will have a blood sample performed for measurement of N-terminal prohormone of B-type natriuretic peptide (NT-proBNP). Patients with an elevated Roche NT-proBNP (≥125 pg/mL) will undergo a transthoracic echocardiogram, clinical examination for signs of HF, HF symptom assessment, an ECG). Patients will undergo echocardiography with a CE-marked, FDA-approved handheld point of care (POC) EchoNous echocardiogram device in all countries. The US2.ai algorithm (which is also CE-marked and FDA-approved) will generate an AI-automated echocardiogram report. In Scotland all patients will also undergo a conventional echocardiogram. Patients who are classified as having heart failure (HFrEF, HFmrEF and HFpEF) will be referred for appropriate follow up.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Routine care arm (No Intervention): Patients in this arm will undergo routine care. They will be managed and followed up as per routine clinical care. They will be remotely monitored for HF events by follow up through electronic records and routinely collected data.
- Investigational arm (Experimental): Patients in this arm will have a blood sample performed for measurement of N-terminal prohormone of B-type natriuretic peptide (NT-proBNP). Patients with an elevated Roche NT-proBNP (≥125 pg/mL) will undergo a transthoracic echocardiogram, clinical examination for signs of HF, HF symptom assessment, an ECG). Patients will undergo echocardiography with a CE-marked, FDA-approved handheld point of care (POC) EchoNous echocardiogram device in all countries. The US2.ai algorithm (which is also CE-marked and FDA-approved) will generate an AI-automated echocardiogram report.
  Interventions: Diagnostic Test: NT-proBNP

INTERVENTIONS:
Diagnostic Test: NT-proBNP — Patients will undergo an NT-proBNP which will guide their future involvement within the study. Patients with an NT-proBNP of ≥125 pg/mL will undergo transthoracic echocardiogram along with a clinical assessment - any diagnosis of HF will result in patients undergoing referral for initiation of guideline directed medical therapy (for HF).
  Arms: Investigational arm

SUMMARY:
This is an international prospective, multicentre, unblinded, randomised-controlled trial. The primary aim is to assess a targeted screening strategy to detect undiagnosed heart failure in high-risk patients.

DETAILED DESCRIPTION:
The primary aim is to assess a targeted screening strategy to detect undiagnosed heart failure (HF) in high-risk patients.

Participants will be recruited from 5-countries (Denmark, Canada, United States of America, Sweden and Scotland). Individual patient data from similar national randomised controlled trials that are independently powered for different efficacy endpoints will be pooled, harmonised and analysed.

After agreeing to consent, patients will be randomised to one of two arms:

"Routine care arm" - patients in this arm will undergo routine care. They will be managed and followed up as per routine clinical care. They will be remotely monitored for HF events by follow up through electronic records and routinely collected data.

OR

"Investigational arm" - patients in this arm will have a blood sample performed for measurement of N-terminal prohormone of B-type natriuretic peptide (NT-proBNP). Patients with an elevated Roche NT-proBNP (≥125 pg/mL) will undergo a transthoracic echocardiogram, clinical examination for signs of HF, HF symptom assessment, an ECG). Patients will undergo echocardiography with a CE-marked, FDA-approved handheld point of care (POC) EchoNous echocardiogram device in all countries. The US2.ai algorithm (which is also CE-marked and FDA-approved) will generate an AI-automated echocardiogram report. In Scotland all patients will also undergo a conventional echocardiogram. Patients who are classified as having heart failure (Heart failure with reduced ejection fraction [HFrEF], Heart failure with moderately reduced ejection fraction [HFmrEF] and Heart failure with preserved ejection fraction [HFpEF]) will be referred for appropriate follow up. In all countries when a handheld echocardiogram reported by AI-automated software does not provide diagnostic images a conventional echocardiogram will be undertaken.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥40 years of age
* Informed consent
* Two or more of the following risk factors for heart failure:

  1. Coronary artery disease (either a previous documented type 1 myocardial infarction or coronary artery bypass grafting or percutaneous coronary intervention or documented stenosis of an epicardial coronary artery [50% left main stem or >70% left anterior descending, circumflex or right coronary artery])
  2. An established diagnosis of diabetes (type 1 or type 2)
  3. Persistent or permanent atrial fibrillation (not paroxysmal atrial fibrillation)
  4. Previous ischemic or embolic stroke
  5. Peripheral arterial disease (previous surgical or percutaneous revascularisation or a documented stenosis greater than 50% of a major peripheral arterial vessel).
  6. Chronic kidney disease (defined as an estimated glomerular filtration rate <60mL/min/1.73m2 or eGFR 60-90mL/min/1.73m2 and UACR >300mg/g).
  7. Regular loop diuretic use (any dose at any dosing interval) for >30 days.
  8. COPD (evidenced by one of the following: PFTs showing airway obstruction, diagnosis by respiratory physician, CT scan reporting presence of emphysema or treatment with national guideline advocated COPD therapy).

Exclusion Criteria:

* Inability to give informed consent e.g., due to significant cognitive impairment
* Previous documented diagnosis of heart failure
* Current renal replacement therapy
* Anyone who, in the investigators' opinion, is not suitable to participate in the trial for other reasons e.g., a diagnosis which may compromise survival over the study period

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3904 (Estimated)
Dates: Start 2022-12-22 (Actual); Primary Completion 2024-06-21 (Estimated); Study Completion 2032-12-21 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of heart failure within 6 months | 6 months

SECONDARY OUTCOMES:
Diagnosis of HFrEF within 6 months | 6 months
People diagnosed with HFrEF receiving GDMT within 6 months | 6 months

OTHER OUTCOMES:
Diagnosis of HFmrEF within 6 months | 6 months
Diagnosis of HFpEF within 6 months | 6 months
People diagnosed with HFmrEF and HFpEF receiving SGLT2i therapy within 6 months | 6 months
Diagnosis of asymptomatic left ventricular dysfunction (LVEF≤40%) within 6 months | 6 months
Time to first heart failure hospitalisation at 1 year | 1 year
Time to first heart failure hospitalisation at 2 years | 2 years
Time to first heart failure hospitalisation at 5 years | 5 years
All-cause mortality at 1 year | 1 year
All-cause mortality at 2 years | 2 years
All-cause mortality at 5 years | 5 years
Time to first occurence of any components of the following clinical composite 1) heart failure hospitalisation 2) all-cause mortality at 1 year | 1 year
Time to first occurence of any components of the following clinical composite 1) heart failure hospitalisation 2) all-cause mortality at 2 years | 2 years
Time to first occurence of any components of the following clinical composite 1) heart failure hospitalisation 2) all-cause mortality at 5 years | 5 years
The incremental cost-effectiveness ratio (ICER) will be expressed as incremental costs/life-year gained | 5 years
The number of patients in the NT-proBNP/echocardiography group with echocardiographic features of potential amyloid as assessed by the US2.ai algorithm report conclusion of "amyloid to be considered" | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mark C Petrie, MbChB, Principal Investigator — University of Glasgow; Carolyn SP Lam, Principal Investigator — Duke-NUS Graduate Medical School
Locations (7):
- Cleveland Clinic, Cleveland, Ohio, United States
- Canada (2):
  - University of British Columbia, Vancouver, British Columbia
  - University of Montreal, Montreal, Quebec
- Rigshospitalet, Copenhagen University Hospital, Copenhagen, Denmark
- Sweden (2):
  - Karolinska University Hospital, Stockholm
  - Uppsala University, Uppsala
- University of Glasgow, Glasgow, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided